CLINICAL TRIAL: NCT02115854
Title: The Value of Labial Biopsy in 65 Patients With Tuberculosis Disease
Brief Title: Labial Biopsy in Patients With Tuberculosis Disease
Status: Completed | Type: Observational
Sponsor: Hopital Lariboisière (Other)
Responsible Party: Principal Investigator, Stephane Mouly, MD PhD, MD PhD, Hopital Lariboisière
Other Study IDs: granuloma1
Record Dates: First submitted 2014-04-10; First posted 2014-04-16 (Estimated); Last update posted 2014-04-16 (Estimated); Status verified 2014-04

CONDITIONS: Tuberculosis; Sarcoidosis
Keywords: usefullness of labial biopsy to distinguish between tuberculosis and sarcoidosis
MeSH Terms: conditions — Tuberculosis; Sarcoidosis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year

GROUPS / COHORTS (1):
- bacteriologically confirmed tuberculosis
  Interventions: Other: labial biopsy

INTERVENTIONS:
Other: labial biopsy

SUMMARY:
The distinction between Tuberculosis disease (TB), a worldwide infective granulomatosis requiring long-term antibiotic treatment, and sarcoïdosis, a rare granulomatous disease successfully treated with high dose steroids is not straightforward and may delay the treatment choice by the physician.

The goal was to evaluate prospectively and consecutively the presence of epithelioid granulomas in salivary glands biopsy of patients with TB.

ELIGIBILITY:
Inclusion Criteria:

* adults above 18 years,
* bacteriologically confirmed tuberculosis

Exclusion Criteria:

* patient not able to sign written consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: bacteriologically confirmed tuberculosis
Sampling Method: Non-Probability Sample
Enrollment: 65 (Actual)
Dates: Start 2010-12; Primary Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
presence of granuloma on labial biopsy | at day zero of treatment of tuberculosis

CONTACTS AND LOCATIONS:
Locations (1):
- Unite de Recherche Thérapeutique, Paris, France